CLINICAL TRIAL: NCT04924049
Title: Video-Assisted Education for Patients With Knee Replacement: Knee Function and Quality of Life
Brief Title: Video-Assisted Education for Patients With Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gulay ALTUN UGRAS, Associate Professor Doctor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mersin University Surgical
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Quality of Life
Keywords: Knee Function; Quality of Life; Surgical Nursing; Video-Assisted Education
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Two-arm [1:1], parallel group, prospective, randomized-controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The video-assisted education group also received routine treatment and care per protocol. Additionally, this patient group watched patient education through video in the patient room before TKR. The contents of the VE were developed by the researchers and included early postoperative care for TKR (knee positioning, early mobilization, pain control, and cold application), ADLs at home (bathing and toileting, eating, sleeping, vehicle driving, housekeeping, sexual life, praying, and maintaining home safety), and gradual exercise at home (for the first 90 days after discharge).
  Interventions: Other: Video-assisted education
- Control (No Intervention): The control group received routine treatment and care per protocol.

INTERVENTIONS:
Other: Video-assisted education — Prior the study, the content and comprehensibility of the VE were evaluated by an orthopedic surgeon, two orthopedic nurses, and a physiotherapist who were not involved in the study and relevant amendments were made based on their suggestions. The preview of the final version of the VE was shown to four patients (10% of the sample) and these patients were excluded from the study. The patients were interviewed by phone calls on a weekly basis and watching VE at home, the frequency of watching VE, and doing home-based exercises were questioned.
  Other Names: Education
  Arms: Experimental

SUMMARY:
Total knee replacement (TKR) is the most effective treatment modality for the correction of knee deformities, increasing the knee functions (KF), relieving pain, and improving quality of life (QoL) of patients. According to the health statistics of the Organisation for Economic Co-operation and Development (OECD), TKR is most commonly used in Sweden (240/100,000), United States (226/100,000), and Austria (215/100,000), while this rate is estimated as 67/100,000 in Turkey (OECD, 2017). Although it has been increasingly applied in Turkey and worldwide, it is associated with postoperative pain, restricted range of motion (ROM), and reduced muscle strength, leading to prolonged recovery process and return to activities of daily living (ADLs) with impaired QoL . In addition, inadequate patient education on knee care and ADLs following TKR may result in repetitive and uncontrollable movements and complications such as severe pain and dislocation. Postoperative complications have been shown to be associated with rehospitalization and redo surgery.

DETAILED DESCRIPTION:
A comprehensive nursing care and patient education are essential to gain independence and return ADLs for patients undergoing TKR. Patient education after TKR increases the success of the operation, improving the healing period, and preventing or minimizing postoperative complications after discharge. All these improve the KF and QoL of the patients. Patients are usually discharged on the first postoperative day, if no complication occurs. Thus, the patient education can be instructed within a very limited period of time, mostly without repetition. Furthermore, patients and/or their relatives may be anxious after TKR and before discharge, leading to difficulties in understanding the education fully or remembering the education given in the hospital. As a result, the use of new technological education tools is inevitable to use the time effectively for nurses.

In recent years, disease-specific video-assisted education (VE) has been increasingly used for patient education. This tool has certain advantages that patients can watch the video repeatedly in every setting, until they understand its content and can remember the content than verbal instructions without limitations of recall memory with decreased anxiety and improved self-care abilities and, eventually, improved patient outcomes . In the present study, we hypothesized that VE could improve the KF and QoL following TKR. Using a holistic approach, we, therefore, aimed to investigate the effect of VE on KF and QoL in patients undergoing TKR.

ELIGIBILITY:
Inclusion Criteria:

Written and verbal consent was obtained to participate in the research,

* 18 years and over,
* Conscious, oriented and cooperative,
* Able to speak and understand Turkish,
* Not diagnosed with any psychiatric illness,
* No known cancer disease,
* Elective surgical intervention applied,
* Total knee replacement applied for the first time,
* Unilateral total knee replacement applied,
* Patients with an Standardized Mini-Mental Test score of 23 and above were included.

Exclusion Criteria:

To research:

* Those who do not agree to participate in the research,
* Under 18 years old,
* Unconscious, without orientation and cooperation,
* Can't speak or understand Turkish,
* Having previously been diagnosed with a psychiatric diagnosis,
* Having a history of cancer,
* Emergency surgical intervention applied,
* Total knee replacement applied before,
* Bilateral (bilateral) total knee replacement applied,
* Patients with an Standardized Mini-Mental Test value below 23 were not included.

Ages: 33 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Physical function will evaluate using Western Ontario and McMaster Universities Osteoarthritis Index | Change from before implementation, after, 1st month and 3rd month
  It consists of a total of 24 items including pain (5 items), stiffness (2 items), and physical function (17 items). Items are rated on a five-point Likert scale as follows: 0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). The highest possible scores which can be obtained are 20 for pain, 8 for stiffness, and 68 for physical function (difficulties experienced when engaging in ADLs). The total score ranges from 0 (the best) to 96 (the worst). Higher scores indicate worse KF, while lower scores indicate better KF.

SECONDARY OUTCOMES:
Quality of life will evaluate using Short Form 36 Quality of Life Scale | Change from before implementation, after, 1st month and 3rd month
  This scale measures eight subscales using 36 self-rating questions including physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. While making the evaluation, a total score is obtained for each subscale separately and these scores are ranges from minimum=0 and maximum=100. Higher scores indicate better quality of life, while lower scores indicate worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Altun Ugras, Doctorate, Study Director — Mersin University
Locations (1):
- Turkey, Mersin University,, Mersin, Turkey/Mersin,Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No